CLINICAL TRIAL: NCT03114007
Title: Inter-Venture: A Cluster Randomized Controlled Trial Investigating the Effect of School-based Personality-targeted Interventions and Collaborative Youth Mental Health Care
Brief Title: Integrated Prevention and Collaborative Care for Youth Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Patricia Conrod, Full professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RBC-CHU-2015
Record Dates: First submitted 2017-03-10; First posted 2017-04-14 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Mental Disorders; Substance-Related Disorders; Quality of Life
Keywords: Mental health problems; Substance misuse; Psychosocial difficulties; Youth
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preventure, Equipe and Inter-Action (Experimental): Preventure program, Equipe program and Inter-Action services: Early personality-targeted interventions for students most at risk of mental health problems and substance misuse (Preventure program), parent program mainly for parents of high risk youth, especially those reporting discord at home (Equipe program) and integrated services for youth with significant internalizing and externalizing problems (Inter-Action services).
  Interventions: Behavioral: Preventure program; Behavioral: Equipe program; Behavioral: Inter-Action services
- Preventure program and Equipe program (Experimental): Early personality-targeted interventions for students most at risk of mental health problems and substance misuse (Preventure program) and parent program mainly for parents of high risk youth, especially those reporting discord at home (Equipe program)
  Interventions: Behavioral: Preventure program; Behavioral: Equipe program
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Preventure program — Personality-targeted interventions conducted using manuals which incorporate psycho-educational, motivational enhancement therapy and cognitive-behavioural components. They include real life 'scenarios' shared by local youth with similar personality profiles. In the first session, participants are guided in a goal-setting exercise, designed to enhance motivation to change behaviour. Psycho-educational strategies are then used to teach participants about the target personality variable and associated problematic coping behaviours like avoidance, interpersonal dependence, aggression, risky behaviours and substance misuse.
  Arms: Preventure program and Equipe program; Preventure, Equipe and Inter-Action
Behavioral: Equipe program — Parent training program designed to be delivered in community settings accessible to large groups of parents of 13 to 18 year olds. It uses a coping modeling problem solving process in which parents are the key players in developing problem solving strategies.
  Parents participate in group workshops with themes related to communication, conflict resolution, cooperative transitions, negotiating, house rules, monitoring, consequences for serious problems and problem solving. Parents are guides to establish solutions to common problems. Readings and videotapes are used in the workshops to guide parents in identifying common challenges in child management, parenting errors, discussing possible consequences and alternative strategies as well as rationales supporting these strategies.
  Arms: Preventure program and Equipe program; Preventure, Equipe and Inter-Action
Behavioral: Inter-Action services — An intervention model designed to provide integrated services for youth with significant symptoms of mental health problems, substance misuse and/or psychosocial difficulties. Young people with such difficulties will benefit from stepped and collaborative care involving interventions of varied intensity adapted to their needs and the severity of their problems. These will include cognitive behavioral therapy, motivational interviews, dialectic behavioral therapy and family interventions provided by multidisciplinary teams of professionals. A case navigator will be in charge of initiating service provision and ensuring a fast and smooth flow of information between indicated services providers.
  Arms: Preventure, Equipe and Inter-Action

SUMMARY:
Mental health problems affect 10-20% of children and adolescents worldwide, with half of affected youth experiencing problems by the age of 14. Despite the early onset of mental health problems, evidence-based prevention and early intervention programs remain scarce. If left untreated, early-onset mental health problems can progress to become severe or chronic conditions, and incur significant medical and societal costs.

The current project proposes an integrated screening and intervention model that was developed involving active youth, family and community engagement. This project, known as Inter-Venture, focuses on reducing barriers to youth mental health care and promoting early screening and intervention by fostering collaboration between school and community-based services providers. The Inter-Venture project is being conducted in the Montreal area (Canada), and consists of three intervention modalities. Namely, 1) systematic school-based screening and personality-targeted interventions for students most at risk of mental health problems and substance misuse (the Preventure program); 2) a parent program designed to strengthen parenting skills and to improve the management of child behavior problems (Cope/EQUIPE program); 3) integrated services provided by a multidisciplinary team of professionals (referred to as Inter-Action) for youth with significant symptoms of mental health problems, substance misuse and/or psychosocial difficulties. The intervention model involves knowledge transfer to boost capacity-building and improve the provision and sustainability of evidence-based interventions in community settings.

The primary goal of the Inter-Venture trial is to assess the potential effect of the school-based targeted interventions and collaborative care in the prevention, early detection and reduction of mental health problems, substance misuse and psychosocial difficulties among young people. The secondary goal is to assess the effect of interventions on school performance and whether the interventions can protect cognitive functions that may be negatively affected by early-onset substance use and mental health problems, and promote cognitive development through the prevention of these difficulties.

DETAILED DESCRIPTION:
The Inter-Venture Trial is a cluster-randomised controlled trial of three intervention modalities developed involving active youth, family and community engagement in the Montreal area: (i) Systematic school-based screening and early personality-targeted interventions for students most at risk of mental health problems and substance misuse (Preventure program); (ii) Community-based parent training program and (iii) Timely and integrated services provided by a multidisciplinary team of professionals (Inter-Action).

The trial will assess the potential effects of some of the components of the intervention model in 45 secondary schools that will be randomly assigned to two intervention conditions (receiving Inter-Action services and the parent training program in addition to Preventure or receiving the Preventure program and the parent training program) and a control arm that will receive treatment as usual. Schools will be matched on their baseline socio-economic status. Approximately 4000 students in participating schools will be invited to complete annual assessments for 5 consecutive years from grade 7 to grade 11.

Based on their scores on the Substance Use Risk Profile Scale, at-risk students will be identified and invited to participate in the Preventure program in the first year of the trial. Parents of grade 7 students reporting discord at home on the Alabama parenting questionnaire will be invited to participate to the parent program. Participating students with clinically significant internalizing and externalizing problems will be invited to receive Inter-Action services. Internalizing and externalizing problems will be assessed using self-report measures such as the Patient Health Questionnaire for Adolescents, the Strengths and Difficulties Questionnaire, the screening tool for the detection of alcohol and drug problems in adolescents (DEP-ADO) and the development and well-being assessment (DAWBA).

Primary outcomes will be the likelihood of reporting a significant level of mental health problems, behavioral problems, substance misuse and poor quality of life among participating youth.

Secondary outcomes will include the severity of the symptoms of mental health and substance use problems, school performance, time to received treatment, time in treatment, quality of care, cognitive functioning and other psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

School inclusion criteria :

- Public or private schools offering regular courses from grade 7 to grade 11.

Student inclusion criteria:

* Being in grade 7 at baseline
* Students' assent to participate
* Parental passive or active consent for students' participation

Parent inclusion criteria

* Being a parent of grade 7 students in a school participating in the parent training program
* Active consent to participate in the study

Exclusion Criteria:

* Schools where the majority of students are coded as special needs students will not be included since the interventions are not adapted to their specific needs

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-09-14 (Estimated); Study Completion 2021-12-14 (Estimated)

PRIMARY OUTCOMES:
Reduced likelihood of having abnormal scores on three scales of the Strength and Difficulties Questionnaire ( conduct problems, emotional problems and hyperactivity scales) at the third and fifth year follow-up. | Annual assessments for 5 years
  The Strengths and Difficulties Questionnaire is a self-report behaviour screening questionnaire used to assess various psychological symptoms and their impact in pediatric populations.
Reduced likelihood of significant alcohol and drug problems at the third and fifth year follow-up assessed by the DEP-ADO, a screening tool for the detection of alcohol and drug problems in adolescents. | Annual assessments for 5 years
  The DEP-ADO is a self-report measure of age of onset, frequency and consequences of alcohol and illicit drug use in adolescents.
Self-reported quality of life at the third and fifth year follow-up assessed by the KIDSCREEN quality of life questionnaire. | Annual assessments for 5 years
  The KIDSCREEN quality of life questionnaire is a self-report measure of four main aspects of adolescents' health-related quality of life: psychosocial functioning, school life, leisure and interpersonal relations.

SECONDARY OUTCOMES:
Reduced likelihood of mental health problems at the third and fifth year follow-up the Patient Health Questionnaire for Adolescents | Annual assessments for 5 years
  The Patient Health Questionnaire for Adolescents is a self-report measure of mental health and behavioral problems such anxiety, depression, and eating disorders among adolescents.
School attendance | Annual assessments for 5 years
  Information on school attendance will be requested from schools
Academic performance | Annual assessments for 5 years
  Grades will be requested to assess academic achievement.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Conrod, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine Research Center, Montreal, Quebec, Canada